CLINICAL TRIAL: NCT02069587
Title: Pomegranate to Reduce Maternal and Fetal Oxidative Stress and to Improve Outcome in Pregnancies Complicated With Preterm Premature Rupture of Membranes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0074-13HYMC
Record Dates: First submitted 2014-02-16; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-01

CONDITIONS: PPROM
Keywords: PPROM; PREGNANCY; POMEGRANATE; OXIDATIVE STRESS
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pomegranate (Experimental): The women in this group will drink pomegranate juice
  Interventions: Dietary Supplement: pomegranate

INTERVENTIONS:
Dietary Supplement: pomegranate
  Other Names: Pomegranate juice

SUMMARY:
Preterm premature rupture of membrane is associated with increased oxidative stress and inflammatory process, enhancing the activity or the availability of antioxidants may modulate the inflammatory response associated with PPROM, thereby reducing oxidative stress and the risk to the fetus. In this study the investigators sought to determine the effects of Pomegranate 1. On the patients (maternal and fetal) oxidative stress and inflammation associated with PPROM. 2. On the time interval from PPROM to delivery and on the patients (fetal )Ph and apger scores

DETAILED DESCRIPTION:
In this study the investigators sought to determine the effects of Pomegranate 1. On the patients (maternal and fetal )oxidative stress and inflammation associated with PPROM. 2. On the time interval from PPROM to delivery and on the patients (fetal )Ph and apger scores

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients
* admitted with PPROM
* between 24-32 weeks of gestation

Exclusion Criteria:

* Women with contractions
* abruption
* monochorionic multiple pregnancy
* abnormal (non-reassuring) cardiotocogram
* meconium-stained amniotic fluid
* signs of intrauterine infection
* major fetal anomalies
* hemolysis
* elevated liver enzymes
* low platelets (HELLP syndrome); or severe preeclampsia.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Maternal and fetal oxidative stress | 10 weeks
  Maternal and fetal oxidative stress will be determined by blood tests.
Maternal and fetal oxidative stress | 10 weeks
  Maternal blood and umbilical cord blodd will be drawn following delivery and oxidative blood markers inflammatory mediators will be assessed

SECONDARY OUTCOMES:
Time interval from PPROM to delivery | 10 weeks
  Time interval from PPROM to delivery, respiratory distress syndrome (RDS), meconium aspiration syndrome, asphyxia, late onset neonatal sepsis, hypoglycemia, necrotizing enterocolitis, hyperbilirubinemia, intraventricular hemorrhage, periventricular leucomalacia, convulsions, other neurological abnormalities, other complications, intrapartum death, total length of hospital stay and admission, and length of stay on neonatal intensive care unit (NICU).
time interval from PPROM to delivery | 10 weeks
  following birth the time interval from PPROM to delivey will be assessed, also RDS, fetal Ph and other neonatal complications

CONTACTS AND LOCATIONS:
Overall Officials: ron beloosesky, Principal Investigator — Hillel Yaffe Medical center technion
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel